CLINICAL TRIAL: NCT06867302
Title: Effectiveness of Single Bolus Versus Continuous Infusion of Dexmedetomidine in Mitigating Agitation in Adults Undergoing Nasal Surgery: a Prospective Randomized Trial
Brief Title: Dexmedetomidine and Agitation After Nasal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Yasser S Mostafa, MD, Lecturer of Anesthesiology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R656
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Nasal Disease; Agitation, Emergence
Keywords: Dexmedetomidine; Emergence agitation; Nasal surgery
MeSH Terms: conditions — Nose Diseases; Emergence Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: the patients will be randomly allocated into two groups based on a computerized randomization table created by a researcher who was not involved in the study. The researcher assigned a random ID to each patient, and a blinded anesthesiologist used this ID while collecting the postoperative data in the surgical ward.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Apart from the anesthesiologists who performed the blocks, all patients, surgeons, and postoperative nurses remained blinded to randomization throughout the study period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolus group (Experimental): single dose 0.5 µg/kg in 15 ml saline over 10 min , started 15 minutes before end of surgery
  Interventions: Drug: Dexmedetomidine in 0.9 % NaCl 1,000 Mcg/250 mL (4 Mcg/mL) INTRAVEN INFUSION BOTTLE (ML)
- Infusion group (Experimental): Infusion of dexmedetomidine at a dose of 0.5 µg/kg/h without loading dose all through intraoperative time
  Interventions: Drug: Dexmedetomidine Injection [Precedex]

INTERVENTIONS:
Drug: Dexmedetomidine in 0.9 % NaCl 1,000 Mcg/250 mL (4 Mcg/mL) INTRAVEN INFUSION BOTTLE (ML) — An infusion given all through intraoperative time
  Other Names: Dexmedetomidine infusion
  Arms: Bolus group
Drug: Dexmedetomidine Injection [Precedex] — Single dose given 15 minutes before end of surgery
  Other Names: Dexmedetomidine bolus
  Arms: Infusion group

SUMMARY:
The main objective of study is to compare dexmedetomidine single bolus dose before extubation with continuous infusion as regards their efficacy in mitigating the incidence of emergence agitation in obese adults undergoing nasal surgery.

DETAILED DESCRIPTION:
Agitation during emergence from general anesthesia is a potentially serious phenomenon that has not been studied in adults as often as in pediatric population. When agitation, serious self-injury, or violence towards the medical team occur, with the risk of aspiration, bleeding, hypoxia, arrhythmias, or simply pulling the endotracheal tubes, removal of drains or catheters. Moreover, agitated patients are not only at risk of developing complications but also, they are labor intensive as they require more medical attention, rescue drugs, and more attending staff till agitation attack safely subside. Recognized risk factors to develop emergence agitation (EA) in adults include ear, nose, and throat surgery, obesity, sevoflurane anesthesia, endotracheal tube, and history of psychological illness. In adults, adjuvants have been co-administered with general anesthesia in order to negate or reduce the incidence of EA especially in patients with identified risk factors.

dexmedetomidine is a highly selective α2 sympatholytic, has been proposed as an attractive candidate for the prophylaxis of EA. By interacting with α2 receptors in locus coeruleus of the pons, Dex exerts its unique anxiolytic, sedative and sympathetic antagonistic action with no respiratory depression. Moreover, it has pain-modulating effect due to interaction with α2 receptor sites in the dorsal horn and supra-spinal regions.

Nevertheless, there have been conflicting data about Dex optimal dose and time of administration when used as prophylaxis against EA. Indeed, different dosing protocols are associated with over sedation, prolonged extubation time, and delayed post-anaesthesia care unit time.

No premedication. Basic general anesthesia monitoring included electrocardiogram, pulse oximetry, non-invasive arterial pressure, and capnography, were recorded every 5 min. Preoxygenation with 100% oxygen for 5 min was performed before fentanyl 1 μg/kg and propofol 1.5-2 mg/ kg, were administered as induction agents. Intubation with facilitated with atracurium besylate 0.5 mg/ kg. The size of endotracheal tubes was 6.5-7.5 mm, for females and males, respectively. Mechanical ventilation was set on 6 ml/kg tidal volume, and respiratory rate was adjusted to keep end-tidal CO2 between 35 and 40 mmHg, in 50% O2/air. All patients at induction were given dexamethasone 4 mg i.v., ondansetron, 4 mg i.v to prevent post-operative nausea and vomiting, plus Ringers lactate solution 6 mg/ kg drip for basic volume maintenance. Blood loss was compensated for with Ringers lactate, intraoperatively. Maintenance of anesthesia was carried out with Isoflurane, regulated at 2-3%, Titrated incremental doses of atropine 0.5 mg, esmolol 10 mg, and ephedrine 6 mg were given i.v., when HR ≤ 45, HR ≥ 120 and MAP ≤ 60, in the mentioned order. ketorolac 30 mg was given I.M., at the time of nasal packing.

When surgery was finished, gentle suction was attempted, non-depolarizing muscle relaxant reverse with atropine, 0.5 mg and neostigmine 0.02 mg/kg was given. Next, isoflurane was turned off and respiration was then converted back to manual ventilation with 100% oxygen at 7 L/min. The patients were not disturbed, except by continual verbal requests to open their eyes. All other stimuli were prevented. Extubation was done when patients were able to breathe spontaneously and interact with verbal demands. When patients were awake, calm, and sedated, they were transferred to the PACU. Patients were discharged from the PACU when their Aldrete score was ≥ 9.

Statistical analysis:

Statistical analysis will be conducted using IBM SPSS Statistics 22 (IBM Corporation, USA). The normal distribution of data will be assessed by the Kolmogorov-Smirnov and Shapiro-Wilk tests. Mean and standard deviation will be used as descriptive statistics for normally distributed numerical variables, while median and interquartile range (25th to 75th percentiles) will be used as descriptive statistics for non-normally distributed numerical variables. In addition, Chi-square test or fisher exact test will be employed to test the significance between categorical variables as appropriate. Independent t test will be employed for numerical data that exhibited normal distribution, whereas the Mann-Whitney test will be used for numerical data that did not adhere to normal distribution. A significance level of p < 0.05 will be deemed to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) Ⅰ or II
* Adults with body mass index (BMI) < 30 Kg/m
* Underwent elective nasal surgery.

Exclusion Criteria:

* Significant comorbidity like hepatic, renal, or cardiac disease
* Auditory impairment
* Cognitive dysfunction
* Substance abuse
* Allergy to the studied medicines
* Planned intensive care admission after the surgery.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Degree of emergence agitation by Richmond Agitation Sedation Scale (RASS) | 5 minutes after operation
  RASS is a 10-point scoring system used to assess patient's level of agitation and sedation: 4 levels for agitation, 1 level for normal (alert and calm), and 5 levels of sedation

SECONDARY OUTCOMES:
Intraoperative heart rate | Every 15 minutes along operation
  Beats / minute
Intraoperative mean arterial blood pressure | Every 15 minutes along operation
  mmHg
Time of first rescue analgesic | 5 minutes before first analgesic request
  in minutes in minutes
Extubation time | 3 minutes after removal of endotracheal tube
  time interval between shutting off anesthetics to extubation (in minutes)
Postanesthesia care unit time | 5 minutes after discharge from recovery unit
  time interval from admission to PACU till patient scored ≥ 9 on Aldrete scale (ready to discharge)
Incidence of use of midazolam | 2 minutes after occurence of emergence agitation
  Yes or no
Numerical rating score (NRS) | Every 10 min in postanesthesia care unit
  10 point scale where zero meaning "no pain" and 10 meaning "the worst pain imaginable"
Total amount of rescue analgesic | 24 hours postoperative
  in milligram
Boezaart Surgical Field Grading Scale | 2 hours intraoperatively
  endoscopically using the six-point score (0-5 Scale) where 0 - No bleeding, 1 - Slight bleeding, no suctioning needed, 2 - Slight bleeding, occasional suctioning needed, 3 - Moderate bleeding, frequent suctioning needed, visibility maintained, 4 - Heavy bleeding, constant suctioning needed, visibility impaired, 5 - Severe bleeding, uncontrolled, surgery impossible
Incidence of bradycardia | 2 hours intraoperatively
  Yes or no
Incidence of hypotension | 2 hours intraoperatively
  Yes or no when mean arterial blood pressure below 60 mmHg
Incidence of nausea | 24 hours postoperative
  Yes or no
Incidence of vomiting | 24 hours postoperative
  Yes or no

OTHER OUTCOMES:
Age | 5 minutes before entering operation department
  in years
Sex | 5 minutes before entering operation department
  Male of female
Weight | 5 minutes before entering operation department
  In kilogram
Height | 5 minutes before entering operation department
  In centimeter
Duration of surgery | 5 minutes after end of surgery
  In minutes

CONTACTS AND LOCATIONS:
Overall Officials: Yasser S Mostafa, MD, Principal Investigator — Fayoum University; Mohamed A Shawky, MD, Study Chair — Fayoum University
Locations (1):
- Fayoum University Hospital, Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu D, Chai W, Sun X, Yao L. Emergence agitation in adults: risk factors in 2,000 patients. Can J Anaesth. 2010 Sep;57(9):843-8. doi: 10.1007/s12630-010-9338-9. Epub 2010 Jun 5. PMID 20526708
- [Background] Hudek K. Emergence delirium: a nursing perspective. AORN J. 2009 Mar;89(3):509-16; quiz 517-9. doi: 10.1016/j.aorn.2008.12.026. PMID 19326585
- [Background] Kim HJ, Kim DK, Kim HY, Kim JK, Choi SW. Risk factors of emergence agitation in adults undergoing general anesthesia for nasal surgery. Clin Exp Otorhinolaryngol. 2015 Mar;8(1):46-51. doi: 10.3342/ceo.2015.8.1.46. Epub 2015 Feb 3. PMID 25729495
- [Background] Lepouse C, Lautner CA, Liu L, Gomis P, Leon A. Emergence delirium in adults in the post-anaesthesia care unit. Br J Anaesth. 2006 Jun;96(6):747-53. doi: 10.1093/bja/ael094. Epub 2006 May 2. PMID 16670111
- [Background] Zhu M, Wang H, Zhu A, Niu K, Wang G. Meta-analysis of dexmedetomidine on emergence agitation and recovery profiles in children after sevoflurane anesthesia: different administration and different dosage. PLoS One. 2015 Apr 13;10(4):e0123728. doi: 10.1371/journal.pone.0123728. eCollection 2015. PMID 25874562